CLINICAL TRIAL: NCT01062984
Title: A Comparison of the Efficacy of Continuous Venovenous Hemofiltration Versus Continuous Venovenous Hemodialysis for Renal Replacement Therapy in Acute Kidney Injury
Brief Title: Continuous Venovenous Hemofiltration Versus Continuous Venovenuous Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: NxStage Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 15947A
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Acute Renal Failure
Keywords: Renal Replacement Therapy
MeSH Terms: conditions — Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Venovenous Hemofiltration (Active Comparator)
  Interventions: Procedure: Continuous Venovenous Hemofiltration (CVVH)
- Continuous Venovenouos Hemodialysis (Active Comparator)
  Interventions: Procedure: Continuous Venovenous Hemodialysis (CVVHD)

INTERVENTIONS:
Procedure: Continuous Venovenous Hemofiltration (CVVH) — The NxStage system will be used for CVVH using the NxStage Cartridge Express dialyzer (polyethersulfone membrane). The blood flow rate will be set at 250 cc/min, and decreased at the discretion of the primary nephrologist's assessment of filter pressures and alarms. Replacement fluid will be delivered pre-filter for CVVH; the target effluent flow rate will be 35ml/kg/hr plus desired ultrafiltration (fluid removal). A maximum of 4.5 L/hr effluent will be prescribed to obese or hypercatabolic patients.
  Arms: Continuous Venovenous Hemofiltration
Procedure: Continuous Venovenous Hemodialysis (CVVHD) — The NxStage system will be used for CVVH and CVVHD using the NxStage Cartridge Express dialyzer (polyethersulfone membrane). The blood flow rate will be set at 250 cc/min, and decreased at the discretion of the primary nephrologist's assessment of filter pressures and alarms. Replacement fluid dialysate will be infused countercurrent to blood flow the target effluent flow rate will be 35ml/kg/hr plus desired ultrafiltration (fluid removal). A maximum of 4.5 L/hr effluent will be prescribed to obese or hypercatabolic patients.
  Arms: Continuous Venovenouos Hemodialysis

SUMMARY:
Acute kidney injury is often treated with the use of continuous renal replacement therapy. Two commonly used treatments are continuous venvenous hemofiltration (CVVH)and continuous venovenous hemodialysis (CVVHD). CVVH uses convective clearance to remove toxins and solutes from the patients circulation, while CVVHD relies on diffusive clearance to remove these same toxins/solutes. This study will evaluate which of these two methods is more effective at clearing the body of waste/solutes.

We hypothesize that renal replacement therapy by either modality (hemodialysis or hemofiltration; CVVHD or CVVH, respectively) using a modern membrane and higher blood flow rates will be associated with similar clearances of both small and middle molecular weight solutes. We further believe that continuous renal replacement therapy using CVVHD will be associated with decreased clotting events and longer hemofilter survival, as well as improved resource utilization (i.e. nursing time, alarms, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older and able to sign consent (or surrogate).
* Must have been referred to the inpatient Nephrology consult service for evaluation of acute kidney injury (AKI).
* Expected survival of at least 48 hours.

Exclusion Criteria:

* Hemoglobin < 8 g/dl
* Serum potassium ≥6.5 milliequivalents per liter (mEq/L)
* Weight > 120kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-01; Primary Completion 2015-09 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
To compare the clearance of urea and creatinine by renal replacement therapy (RRT) using continuous venovenous hemofiltration versus continuous venovenous hemodialysis. | 48 hours

SECONDARY OUTCOMES:
To compare the clearance cystatin C and inflammatory cytokines (IL-6 and IL-10) by RRT using continuous venovenous hemofiltration versus continuous venovenous hemodialysis. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jay Koyner, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356